CLINICAL TRIAL: NCT04916600
Title: NET Device as a Non-Pharmacological Alternative to Medication for Opioid Withdrawal Symptom Reduction and Abstinence
Brief Title: NET Device for Treating Opioid Use Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: NET Recovery Corp (Unknown); Isaiah House (Unknown)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Professor of Psychiatry and Behavioral Neurosciences; and Director, Substance Addiction Research Division, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 21-07-3820
Record Dates: First submitted 2021-06-03; First posted 2021-06-07 (Actual); Results first posted 2025-08-07 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This study is prospective, randomized, double-blind, parallel-group, sham-controlled and superiority in design. Study enrollees will be assigned in equal proportions (1:1) to one of two groups: active or sham treatment. Group assignment will be stratified by sex. The biostatistician will perform stratified randomization to maintain balance between active and sham groups. The biostatistician will maintain the blinding so that the study sponsor, PI, study monitor, research assistants, treatment staff, and the participants remain blinded. No interim analysis is planned.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sham controls for placebo effects, and is designed to minimize sham recognition by participants, research, and treatment personnel. Active and sham arms will receive identical device care and use instructions, equipment, and attachment locations. Visual cues from the device "heartbeat" indicator (light-emitting diode) indicate the device is working. Sham and active both use the NET device without alteration. Sham uses a lead wire rendered non-conductive beforehand, preventing electrical stimulation. The biostatistician will randomly and uniquely assign a pre-printed Study Device Number (SDN) to each lead wire by overlaying a heat shrink tube, pre-printed with a unique SDN, recording the active and sham assignments. Lead wires are inserted into the device. The biostatistician will keep the data in a secure database and will not be involved in recruitment or study procedures. Unblinding will only occur when necessary for treating an adverse event.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- NET active (Experimental): Active, non-invasive, alternating current transcutaneous stimulation through electrodes placed transcranially on the mastoid regions. Treatment is self-administered, with participant control of device output level and duration according to perceived benefit. Minimum treatment duration is one-hour, with self-administered extension not to exceed 7 days.
  Interventions: Device: NET
- NET sham (Sham Comparator): Sham, non-invasive, stimulation through electrodes placed transcranially on the mastoid regions. Treatment is self-administered, with participant control of device output level and duration according to perceived benefit. Minimum treatment duration is one-hour, with self-administered extension not to exceed 7 days.
  Interventions: Device: NET

INTERVENTIONS:
Device: NET — NET is an investigational device that received CE-Mark in April 2009 as a Class IIa active medical device

SUMMARY:
This prospective, randomized, double-blind, parallel-group, sham-controlled, superiority study will evaluate the effectiveness of the NET Device in treating persons with Opioid Use Disorder (OUD) without use of Medications for OUD (MOUD) for persons who have expressed a desire to be opioid abstinent without use of MOUD.

DETAILED DESCRIPTION:
The primary study objective is to determine whether use of the active NET Device produces a clinically meaningful decrease in opioid withdrawal symptom severity from baseline to 1-hour in persons with OUD experiencing moderate or greater symptoms of opioid withdrawal.

The NET Device is an investigational Non-Significant Risk device that delivers alternating current via surface electrodes placed transcranially on the mastoid regions. All participants will be screened and undergo evaluation at Isaiah House, a treatment center located in Willisburg, KY. Individual participant treatment (duration of the active/sham device use) is 1 hour and extendable by participant choice, but not to exceed 7 days, delivered at the inpatient facility (typically 28 days duration), with weekly follow-up assessments (efficacy and safety endpoints) following discharge (by video) for a 12-week outpatient study period. Total elapsed time will typically be 16 weeks.

The primary study endpoint is a clinically meaningful decline in COWS total score (defined as a ≥15% reduction) from baseline to 1-hour after start of active NET stimulation.

The first secondary endpoint is a comparison of the decrease in COWS total scores from baseline to 1-hour after start of intervention for active vs sham.

The second secondary efficacy endpoint is a comparison of the percentage of weeks of abstinence from illicit opioid use without the use of MOUD for active vs sham over 12 outpatient weeks following discharge from residential care.

The secondary safety endpoint is the prevalence of all adverse events (AEs) and serious adverse events (SAEs) assessed from day 1 baseline to the end of study, and adverse device effects (ADEs), serious adverse device effects (SADEs), unanticipated adverse device effects (UADEs), and device deficiencies assessed from day 1 baseline to end of day 7.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study (including inpatient stay and participation in video assessments and remote drug screens for the duration of the 12-week outpatient study period).
3. Stated desire to be opioid abstinent without medications for treating opioid use disorder.
4. Male or female, aged 18-65 years.
5. In good general health as evidenced by medical history.
6. Meet Diagnostic and Statistical Manual (DSM)-5 criteria for opioid use disorder (any severity level) alone or comorbid with stable medical diseases (except for certain medications below).
7. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method for the duration of the study.
8. Initiating opioid discontinuation at Isaiah House.
9. Clinical Opiate Withdrawal Scale (COWS) total score is 13 or greater.

Exclusion Criteria:

1. Acute/unstable illness: conditions making it unsafe to participate.
2. Chronic illnesses: primarily seizures and dementing illnesses, including medications for these neurological conditions.
3. Current serious psychiatric disease: psychosis, bipolar disorder.
4. Requiring detoxification from alcohol or benzodiazepines.
5. Current use of anxiolytics, hypnotics (prescription and over the counter), antidepressants, anticonvulsants, sedating histamine-1 receptor subtype antihistamines (non-sedating second generation histamine-4 receptor subtype antihistamines are allowed), prescription and over the counter stimulants.
6. Current diagnosis other than opioid use disorder requiring chronic opioid treatment.
7. Presence of a cardiac pacemaker.
8. Pregnancy or lactation. Females who do not agree to sexual abstinence or are heterosexually active and not using (self-report) medically approved birth control measures (sterilization, tubal ligation, oral/depot contraceptives, abstinence, intrauterine device, barrier method such as condom/foam, or a cervical cap combined with a spermicide), are not eligible.
9. Receiving extended-release buprenorphine (Sublocade) within 300 days of enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mark K Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Isaiah House Treatment Center, Willisburg, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
This is a proprietary device and company-sponsored clinical trial. No IPD will be made available.

REFERENCES:
- [Result] Greenwald MK, Ghosh S, Winston JR. A randomized, sham-controlled, quintuple-blinded trial to evaluate the NET device as an alternative to medication for promoting opioid abstinence. Contemp Clin Trials Commun. 2022 Oct 18;30:101018. doi: 10.1016/j.conctc.2022.101018. eCollection 2022 Dec. PMID 36303593
- [Result] Greenwald MK, Arfken CL, Winston JR. A randomized, sham-controlled clinical trial to evaluate the NET Device for reducing withdrawal symptom severity during opioid discontinuation. Front Psychiatry. 2025 Feb 19;16:1510428. doi: 10.3389/fpsyt.2025.1510428. eCollection 2025. PMID 40046990
- [Derived] Greenwald MK, Arfken CL, Winston JR. Post-discharge use of opioids, psychostimulants, and treatment medications following residential opioid discontinuation with NET Device monotherapy. Front Psychiatry. 2025 Oct 15;16:1627267. doi: 10.3389/fpsyt.2025.1627267. eCollection 2025. PMID 41169495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 108 participants were enrolled. 53 were enrolled in the active device arm and 55 were enrolled in the sham device arm.
Pre-assignment Details: Randomization to active vs. sham conditions was preserved.
Period: Overall Study
Arm/Group | NET Active | NET Sham
Started | 53 | 55
Completed | 53 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NET Active | NET Sham | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (7.6) | 33.4 (9.1) | 34.1 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 31 | 33 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 51 | 52 | 103
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 48 | 49 | 97
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 53 | 55 | 108

OUTCOME MEASURES:

1. Primary Outcome: Clinically Meaningful Decrease in Opioid Withdrawal Symptom Severity
Description: percentage of participants with 15% or greater reduction (from baseline to 1 hour device utilization) in total score on the Clinical Opiate Withdrawal Scale (COWS); scores range from 0 to 48, with higher scores indicating more severe withdrawal
Time Frame: from baseline to 1-hour of device stimulation
Population: All enrolled participants who completed 1 hour of randomly assigned intervention (active or sham)
Measure: Number; unit: percentage of participants
Arm/Group | NET Active | NET Sham
Number analyzed (Participants) | 53 | 55
percentage of participants | 98.1 | 83.6

2. Secondary Outcome: Comparison of Change in Opioid Withdrawal Symptom Severity Between Active and Sham Device Treatment
Description: Difference in percentage change in total score on the Clinical Opiate Withdrawal Scale (COWS) between active and sham groups; scores range from 0 to 48, with higher scores indicating more severe withdrawal
Time Frame: from baseline to 1-hour of device stimulation
Population: All enrolled participants who completed 1 hour of randomly assigned device utilization (active or sham)
Measure: Mean (Standard Deviation); unit: percentage change in COWS score
Arm/Group | NET Active | NET Sham
Number analyzed (Participants) | 53 | 55
percentage change in COWS score | -61.7 (4.9) | -45.8 (8.9)

3. Secondary Outcome: Comparison of the Rate of Illicit Opioid Abstinence Without Medications for Treating Opioid Use Disorder
Description: Percentage of participants with no illicit opioid use without use of medications for treating opioid use disorder (based on weekly post-discharge timeline followback interview). This outcome definition is a conjunction (i.e. required combination) of a participant not using any illicit opioid AND not using any medication for treating opioid use disorder at each assessment time point. This is consistent with the intent of the study to examine the efficacy of the device as a monotherapy (without relying on medications).
Time Frame: Overall percentage of zero use-days (no illicit opioids without medications for treating opioid use disorder) during post-discharge weeks 1-12
Population: All participants who (during the inpatient period) received randomly assigned device exposure (active or sham)
Measure: Number; unit: percentage of participants
Groups:
- Active Device >=24 Hour Utilization: Those randomly assigned to active device who self-administered stimulation >= 24 hours
- Active Device <24 Hours Utilization: Those randomly assigned to active device who self-administered stimulation <24 hours
- Sham Device >= 24 Hours: Those randomly assigned to sham device who self-administered stimulation >=24 hours
- Sham Device <24 Hours Utilization: Those randomly assigned to sham device who self-administered stimulation <24 hours
Arm/Group | Active Device >=24 Hour Utilization | Active Device <24 Hours Utilization | Sham Device >= 24 Hours | Sham Device <24 Hours Utilization
Number analyzed (Participants) | 23 | 25 | 21 | 34
percentage of participants | 87.0 | 40.0 | 52.4 | 52.9

4. Secondary Outcome: Rate of Adverse Events
Description: All adverse events including dermal rash, inflammation, or other adverse events from use of the device
Time Frame: Number of adverse events during inpatient device use (which can range across participants from 1 hour to 7 days)
Population: All participants receiving exposure to the randomly assigned intervention (active or sham)
Measure: Count of Participants; unit: Participants
Arm/Group | NET Active | NET Sham
Number analyzed (Participants) | 53 | 55
Participants | 1 | 0

5. Post Hoc Outcome: Zero Days Use
Description: Percentage of participants with zero days of using illicit opioids, illicit psychostimulants, and medications for treating opioid use disorder (MOUD)
Time Frame: Days 1 to 30 post-discharge
Measure: Number; unit: percentage of participants
Groups:
- Active Device Use >=24 Hours: Participants randomly assigned to receive active NET Device, who self-administered stimulation for 24 hours or more.
- All Other Participants: Participants randomly assigned to active NET Device who self-administered stimulation <24 hours, and participants randomly assigned to the sham device (regardless of duration of self-administration)
Arm/Group | Active Device Use >=24 Hours | All Other Participants
Number analyzed (Participants) | 23 | 80
percentage of participants | 87.0 | 65.0
Statistical Analysis 1: Comparison: Active Device Use >=24 Hours vs All Other Participants; Test type: Superiority; p = .043, Chi-squared — The threshold for statistical significance was p = .05; Difference in percentages = 22.0 — Treatment difference = Active device >=24 hour group - remainder of participants (Active <24 hr, Sham >=24 hr, and Sham <24 hr groups)

6. Post Hoc Outcome: Average Number of Use-days
Description: Average number of days using illicit opioids, illicit psychostimulants, or medications for opioid use disorder (MOUD)
Time Frame: Days 1 to 30 post-discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Active Device Use >=24 Hours | All Other Participants
Number analyzed (Participants) | 23 | 80
days | 0.5 (1.9) | 3.9 (7.6)
Statistical Analysis 1: Comparison: Active Device Use >=24 Hours vs All Other Participants; Test type: Superiority; p = .032, t-test, 2 sided — The threshold for statistical significance was p = .05; df=101; Mean Difference (Net) = -3.4

ADVERSE EVENTS:
Time Frame: Daily from the time of initiating device use (inpatient day 1) throughout the remaining inpatient period (up to 28 days), and continuing weekly from post-discharge week 1 throughout the end of the post-discharge period (end of week 12).
Description: AEs were queried systematically throughout the inpatient period and weekly during the post-discharge period.
Arm/Group | NET Active | NET Sham
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/55
Other Adverse Events (participants affected / at risk) | 1/53 | 0/55
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NET Active (N=53) | NET Sham (N=55)
Headache (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT04916600/Prot_SAP_001.pdf